CLINICAL TRIAL: NCT05533216
Title: Upper Limb Functional Testing in Athletes: Elaboration of Normative Data
Brief Title: Upper Limb Functional Testing in Athletes
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Physiotherapist, University of Liege
Other Study IDs: UL functional testing
Record Dates: First submitted 2022-08-29; First posted 2022-09-08 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Functional Performance
Keywords: prevention; performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Performance of different upper limb functional tests — The participants will have to perform 3 to 5 different upper libm functional tests, depends on the sport they practice.

SUMMARY:
The aim of this study is to elaborate sports-specific normative data for different upper limb functional tests.

About 250 sportspeople, aged between 14 and 35 years, and practicing an upper limb sport, will be recruited. They will performed some of the following tests, based on the sport they practice :

* Upper Quarter Y Balance Test
* Athletic Shoulder Test
* Single Arm Medicine Ball Throw
* Countermovement push-ups
* Closed Kinetic Chain Upper Extremity Stability Test
* Upper Limb Rotation Test
* Posterior Shoulder Endurance Test
* Seated Shot Put Test

ELIGIBILITY:
Inclusion Criteria:

* To practice an upper limb sport, at least 5 or 6 hours a week

Exclusion Criteria:

* Shoulder pain, injury or surgery during the last 6 months

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The participants will have to practice an upper limb sport for, at least, 3 years and with a volume of at least 5-6 hours a week.
Sampling Method: Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Score Upper Quarter Y Balance Test | through study completion
  the maximal distance, in centimeters, will be measured
Athletic Shoulder Test | through study completion
  maximal peak force, in Newton, will be measured, using a handheld dynamometer
Single Arm Medicine Ball Throw | through study completion
  maximal distance, in meters, will be measured
Closed Kinetic Chain Upper Extremity Stability Test | through study completion
  the maximal number of touches, in 15 seconds, will be measured
Upper Limb Rotation Test | a single measurement
  the maximal number of touches, in 15 seconds, will be measured
Posterior Shoulder Endurance Test | through study completion
  time until exhaustion (in seconds)
Seated Single Arm Shot Put Test | through study completion
  maximal distance, in meters, will be measured
Shoulder rotators isometric strength | through study completion
  maximal peak force will be measured in Newton, using a handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Camille Tooth, Principal Investigator — University of Liege
Locations (1):
- University of Liège, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided